CLINICAL TRIAL: NCT01255423
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Sodium Topical Gel (DSG) 1% Applied 4 Times Daily in Subjects With Acute Ankle Sprain
Brief Title: Efficacy and Safety of Diclofenac Sodium Topical Gel 1% Applied 4 Times Daily in Subjects With Acute Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197-P-320
Record Dates: First submitted 2010-12-01; First posted 2010-12-07 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Ankle Sprain
Keywords: Ankle sprain, soft tissue injury
MeSH Terms: conditions — Ankle Injuries; Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac sodium topical gel 1% (Experimental)
  Interventions: Drug: Diclofenac sodium topical gel 1%
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac sodium topical gel 1% — Diclofenac sodium topical gel 1%, 4 times daily
  Arms: Diclofenac sodium topical gel 1%
Drug: Placebo — Placebo, 4 times daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Diclofenac Sodium Topical (DSG) 1% compared with placebo applied four times a day in subjects with acute ankle sprains under 'in-use' conditions, in particular with regard to pain relief.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged 18 years and over.
2. Acute sprain of the lateral ankle, Grade I-II, meeting baseline pain intensity level.
3. Injury within past 12 hours.

Exclusion criteria:

1. Pain medication was taken within the 6 hours that precede randomization.
2. During the past 3 months: Grade I-III sprain of the same ankle.
3. During the past 6 months: Grade II-III sprain, any other significant injury (such as fracture or torn ligament), or surgery (except for skin or nails) of the same ankle or foot.
4. Pain or instability in the same ankle attributable to previous ankle sprain or any other trauma.
5. Ankle sprain attributable to a known disease affecting the ligaments, such as ligament hyperlaxity due to connective tissue disease (e.g., Marfan's syndrome, Down's syndrome, Ehlers-Danlos syndrome).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis
Locations (9):
- United States (9):
  - Birmingham, Alabama
  - Aventura, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Berlin, New Jersey
  - Columbia, South Carolina
  - El Paso, Texas
  - Houston, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start 30 Nov 2010 Study end 17 Juin 2011
Period: Overall Study
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Started | 104 | 102
Completed | 101 | 99
Not Completed | 3 | 3
Not completed — Abnormal Laboratory value | 3 | 2
Not completed — Use of prohibited medications | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo | Total
Number analyzed (Participants) | 104 | 102 | 206
Age Continuous [Mean (Standard Deviation); unit: years] | 31.0 (13.1) | 30.8 (13.9) | 30.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 57 | 119
  Male | 42 | 45 | 87
Region of Enrollment [Number; unit: participants]
  United States | 104 | 102 | 206
18 years and above [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  18 years and above | 104 | 102 | 206

OUTCOME MEASURES:

1. Primary Outcome: Pain on Movement
Description: Pain on movement at 72 hours assessed on a 100 mm visual analog scale with anchors at 0= "No pain" and 100= "Extreme pain"
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 102
mm | 37.4 (25.2) | 38.8 (24.1)

2. Secondary Outcome: Pain on Movement
Description: Pain on movement at 24 hours and 7 days assessed on a 100 mm visual analog scale with anchors at 0= "No pain" and 100= "Extreme pain"
Time Frame: 24 hours and 7 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 102
mm
  24 hours | 52.9 (22.5) | 53.1 (22.6)
  7 days | 19.4 (23.1) | 22 (23.5)

3. Secondary Outcome: Onset of Pain Relief
Description: Onset of perceptible pain relief
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Hour
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 102
Hour | 2 [2 to 2.2] | 2 [1.8 to 6.0]

4. Secondary Outcome: Tenderness
Description: Tenderness at 24 and 72 hours and 7 days. Change from baseline. Tenderness was measured by a calibrated algometer in order to quantify the pressure pain threshold, a measure of tenderness.
Time Frame: Change from baseline at 24 and 72 hours, 7 days
Measure: Mean (Standard Deviation); unit: N/cm^2
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 102
N/cm^2
  Change from baseline at 24 Hours | 2.3 (8.2) | 1.3 (7.7)
  Change from baseline at 72 Hours | 6.4 (11.9) | 5.5 (11.4)
  Change from baseline at 7 Days | 12.1 (13.3) | 11.9 (10.6)

5. Secondary Outcome: Ankle Joint Function
Description: Ankle joint function score (Karlsson Scoring scale which ranges from 0 "worst possible score" to 90 "best possible score")at 24 and 72 hours and 7 days.
Time Frame: 24 and 72 hours, 7 days
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Number analyzed (Participants) | 104 | 102
Total score
  24 Hours | 30.1 (18.7) | 30.7 (17.6)
  72 Hours | 47.2 (19.3) | 46.1 (19.8)
  7 days | 68.8 (20.0) | 66.4 (21.5)

ADVERSE EVENTS:
Arm/Group | Diclofenac Sodium Topical Gel 1% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/102
Other Adverse Events (participants affected / at risk) | 11/104 | 8/102
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Topical Gel 1% (N=104) | Placebo (N=102)
Nervous Sytem disorders (Nervous system disorders) | 5 (5) | 3 (3)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Infection and infestations (Infections and infestations) | 2 (2) | 0 (0)
General disorders and administration site conditions (General disorders) | 1 (1) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Injury poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator